CLINICAL TRIAL: NCT05927636
Title: Systemic Treatment Related Toxicity Identified With a Smartphone APPlication Measuring Step Count - Prospective Cohort Study
Brief Title: Systemic Treatment Related Toxicity Identified With a Smartphone APPlication Measuring Step Count
Acronym: STAPPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Medisch Centrum Leeuwarden (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-13469
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Systemic Treatment; Physical Activity; Toxicity Due to Chemotherapy
Keywords: Cancer; Systemic treatment; Toxicity; Physical activity; Smartphone; wearable; Daily step count
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients with cancer referred for systemic treatment of the outpatient clinic at the departments of Medical Oncology at participating centres.

SUMMARY:
The goal of this observational study is to investigate whether daily physical activities measured with a smartphone are related to the possible side effects or other physical complaints that arise as a result of cancer treatment. The investigators want to test whether the number of steps per day, both before and during treatment, are related to possible side effects or other physical complaints of the treatment using a smartphone. Knowledge about this relationship gives us possible starting points to prevent and/or reduce side effects and improve treatment outcomes. Additional research would then be needed.

The investigators also want to investigate whether these daily measurements are feasible for patients undergoing treatment.

Participation in the study involves measuring daily physical activity from the week before treatment until the first 3 months of treatment have been completed. This is done by tracking daily steps with patients own phone using the OncoSTAPP application.

DETAILED DESCRIPTION:
Rationale: Systemic treatment of patients with cancer has a multimodal approach with the goal of balancing quantity and quality of life. Treatment decisions are influenced by tumour and patient-related characteristics. Additionally, in clinical practice performance status is used to identify whether a patient is sufficiently fit for systemic treatment, as it has shown to be a valid prognostic factor for survival and adverse events during treatment. However, treatment-related toxicities and hospitalisations occur frequently during systemic treatment.

The disadvantages of performance status assessed with ECOG or Karnofsky, is that it is a subjective measurement which is prone to bias and has high interobserver variability. Also a patient's self-reported physical function is significantly associated with shorter (progression-free) survival, but it is also subjective and is prone to multiple forms of bias. Objective assessment of physical function might be a good alternative to counteract these shortcomings. A higher level of physical activity is associated with a reduction in cancer specific mortality and can be measured with accelerometers, pedometers or multisenor systems like smartphones.

Wearable measured step count assessed with a wrist worn device provided by the investigators has shown to be associated with adverse events. However, these devices cannot be provided to all patients in clinical practice.

Recently, the investigators showed that the smartphones' assessments of physical activity (step count), have excellent agreement with accelerometer assessments of physical activity and good test-retest reliability. Furthermore this smartphone measurements were associated with early trial discontinuation in phase 1/2 cancer trials.

The investigators hypothesize that a low baseline and/or a reduction in physical activity (step count) measured with smartphones will be predictive for clinically relevant adverse events during systemic treatment. Adding objective information of physical function in the process of selecting the best treatment for a patient may help prevent unnecessary adverse events. Additionally, a detection of a decline in physical activity during treatment may identify upcoming adverse events early, allowing timely management/support. This may help to optimize treatment and quality of life.

Objective: Primary objectives: 1) To determine whether baseline physical activity, measured by the number of steps per day with a smartphone, is associated with clinically relevant adverse events during treatment.

2) To determine whether changes in physical activity, measured by the number of steps per day with a smartphone, are associated with clinically relevant adverse events during treatment.

Clinically relevant adverse events during treatment are defined as hospitalizations, early treatment discontinuation, relative dose intensity below 70% and mortality.

Secondary: Patients' acceptability of the application. The association of physical activity with relative dose intensity, progression free and overall survival. The association between the oncologists' estimates and clinically relevant adverse events during treatment, and the possible added value of objective assessments of physical activity.

Study design: Prospective observational cohort study.

Study population: 411 patients with cancer referred for systemic treatment at the departments of Medical Oncology at participating centres.

Intervention: N/A.

Main study parameters/endpoints: Collection of daily number of steps will start in the week before treatment and will continue for the first 3 months of systemic treatment. Mean number of steps per day will be measured passively with a smartphone application on patients' own smartphones. Primary endpoint is any clinically relevant adverse events during treatment, defined as hospitalizations, significant dose modifications of treatment and mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in this study will not cause any additional risks or expected benefits for participants. No extra visits to the hospital will be necessary. It will provide us knowledge, which may be used in the future to better select patients for systemic treatment.

Patients will be asked to carry their smartphone on them during the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of cancer with an indication of starting systemic treatment
* Knowledge how to handle smartphone with iOS version 11 or higher or Android version 7.0 or higher.
* Mastery of Dutch language
* Able and willing to give written informed consent

Exclusion Criteria:

* Cognitive disorders or severe emotional instability
* Wheelchair-depended at home, or immobile due to for example fracture
* Already participating in an exercise trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with cancer referred for systemic treatment of the outpatient clinic at the departments of Medical Oncology at participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | From enrollment to the end of observation period (90 days on systemic treatment)
  Mean number of steps per day measured with a smartphone. At baseline and during treatment
Number of patients with a hospitalization | From enrollment to the end of observation period (90 days on systemic treatment)
  Hospitalizations during treatment related to the therapy; will be combined into Clinically relevant adverse events during treatment
Number of patients with a treatment discontinuation | From enrollment to the end of observation period (90 days on systemic treatment)
  Early treatment discontinuation, within the first 3 months; will be combined into Clinically relevant adverse events during treatment
Number of patients with a RDI <70% | From enrollment to the end of observation period (90 days on systemic treatment)
  Relative dose intensity (RDI) below 70%; will be combined into Clinically relevant adverse events during treatment
Rate of mortality | From enrollment to the end of observation period (90 days on systemic treatment)
  Mortality due to treatment toxicity; will be combined into Clinically relevant adverse events during treatment
Relative dose intensity (RDI) of systemic treatment | From enrollment to the end of observation period (90 days on systemic treatment)
  The percentage of planted dose and time between doses will be retrieved form patients' medical records (EPIC). The RDI will be calculated by total percentage of given dose divided by the proportion of the actual time in relation to the standard time. RDI=(Total percentage of given dose)/((Actual time)/(Standard time))*100

SECONDARY OUTCOMES:
Physician's rated performance status | At enrollment
  The Eastern Cooperative Oncology Group/World Health Organization Performance Status (ECOG/WHO-PS) will be determined by the treating physician before treatment as stated in the current treatment guidelines of the departments of Medical Oncology. scale 0 to 5, with 0 denoting perfect health and 5 death.
Oncologists' estimates of high toxicity risk during treatment | At enrollment
  Question if patients are defined as at high (>50%) or low risk of dose limiting (>25% or discontinuation) toxicity during the first 3 months of systemic treatment. This will be documented in patients' medical records (e.g. EPIC).
Overall survival | From enrollment until the date of death from any cause, assessed up to 2 years
  Overall survival is defined as the time between start of trial participation and death of any cause and will be tracked via the patients' medical records (e.g. EPIC).
Progression free survival | From enrollment until the date of first documented progression assessed up to 2 years
  Progression free survival is defined as the time between start of systemic treatment and the clinically or radiologically confirmation of progressive disease (established via RECIST-criteria) and will be tracked via the patients' medical records (e.g. EPIC).
Proportion of patients with correctly collected data | From enrollment to the end of observation period (90 days on systemic treatment)
  Validity of the smartphone application will be assesed by the proportion of patients correctly collected the data.
Patients experience with smartphone application | At the end of the observation period (90 days on systemic treatment), or reported spontaniously by the patient
  A consecutive sample of patients will be contacted for a short interview about the use of the smartphone application, until data saturation. Any spontaneously reported reactions about the smartphone application will be collected.

OTHER OUTCOMES:
Patient characteristics, age | at enrolement
  age at enrolement, in years
Patient characteristics, weight | at enrolement
  body weight, in kilograms
Patient characteristics, heigth | at enrolement
  height, in meters
Patient characteristics, comorbidities | at enrolement
  Comorbidities of the patiënt, with the Charlson Comorbidity Index (CCI)
Patient characteristics, tumour | at enrolement
  tumour type and stage, pathology findings.
Patient characteristics, previous treatment | at enrolement
  previous treatments related to current tumour. including surgery, radiotherapy and all systemic treatments
Patient characteristics, treatment | at enrolement
  treatment characteristics, type of systemic treatment
Patient characteristics, number of medication | at enrolement
  Total number of medications before current systemic treatment.
Patient characteristics, Hemoglobin | at enrolement
  laboratory finding captured as routine care at enrolement, Hemoglobin (mmol/L)
Patient characteristics, Leukocytes | at enrolement
  laboratory finding captured as routine care at enrolement, Leukocytes (10**09/L)
Patient characteristics, Trombocytes | at enrolement
  laboratory finding captured as routine care at enrolement, Trombocytes (10**09/L)
Patient characteristics, Neutrophils | at enrolement
  laboratory finding captured as routine care at enrolement, Neutrophils (10**09/L)
Patient characteristics, Lymphocytes | at enrolement
  laboratory finding captured as routine care at enrolement, Lymphocytes (10**09/L)
Patient characteristics, Sodium | at enrolement
  laboratory finding captured as routine care at enrolement, Sodium (mmol/L)
Patient characteristics, Urea | at enrolement
  laboratory finding captured as routine care at enrolement, Urea (mmol/L)
Patient characteristics, Creatinine | at enrolement
  laboratory finding captured as routine care at enrolement, Creatinine (umol/L)
Patient characteristics, Creatinine clearance | at enrolement
  laboratory finding captured as routine care at enrolement, Creatinine clearance (ml/min/1.73m2) CKD-EPI-GFR
Patient characteristics, Alanine aminotransferase | at enrolement
  laboratory finding captured as routine care at enrolement, alanine aminotransferase (U/L) (ALAT)
Patient characteristics, Aspartate aminotransferase | at enrolement
  laboratory finding captured as routine care at enrolement, Aspartate aminotransferase (U/L) (ASAT)
Patient characteristics, Serum Lactate Dehydrogenase | at enrolement
  laboratory finding captured as routine care at enrolement, Serum Lactate Dehydrogenase (U/L) (LDH)
Patient characteristics, Alkaline phosphatase | at enrolement
  laboratory finding captured as routine care at enrolement, Alkaline phosphatase (U/L)
Patient characteristics, Serum Albumin | at enrolement
  laboratory finding captured as routine care at enrolement, Serum Albumin (g/L)
Patient characteristics, C-reactive protein | at enrolement
  laboratory finding captured as routine care at enrolement, C-reactive protein (mg/L)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Erasmus MC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
No current plans for data sharing. Patients gave informed consent to share data with studies in line with the current research question. Data availible on request.
Time Frame: Till 15 years from start data collection
Access Criteria: Research question in line with current

REFERENCES:
- See also: Website with patient information in dutch — https://www.radboudumc.nl/lopende-onderzoeken/stapps